CLINICAL TRIAL: NCT00386412
Title: Phase II, Multicentric, Prospective and Opened Clinical Trial of Advance Valganciclovir Treatment of CMV in Allogenic Hematopoietic Progenitors Transplant
Brief Title: TAMOVALCIR in Allogenic Hematopoietic Progenitors Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Pethema, pethema
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-002813-19.; TAMOVALCIR in alogenic
Record Dates: First submitted 2006-10-09; First posted 2006-10-11 (Estimated); Last update posted 2009-09-18 (Estimated); Status verified 2009-09

CONDITIONS: Cytomegalovirus Infection
Keywords: Cytomegalovirus infection
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Valganciclovir

INTERVENTIONS:
Drug: Valganciclovir — 900 mg/ 12 h oral, 2 weeks 900 mg/ 24 h oral, 2 weeks

SUMMARY:
PRINCIPAL ENDPOINT To value valganciclovir efficacy in advance treatment of CMV in patients received allogenic transplant with a uniform treatment.

SECONDARY ENDPOINT To value valganciclovir security in advance treatment of CMV in in patients received allogenic transplant with a uniform treatment.

The security will be valued by the % of patients that:

Will have negative CMV Neutropenia <1000 neutrophils/mm3 or <500 neutrophils/mm3 in the first 35 days of treatment - follow-up Renal toxicity in the first 35 days of treatment - follow-up (defined by elevated creatinine >1mg/dL or twice the basal value) CMV illness during the treatment or in the next 2 months Blood Antigenemia / PCR positive in the next 2months of treatment

This dates Hill be compared with a patients control group treated with intravenous valganciclovir

DETAILED DESCRIPTION:
Clinical trial with a drug in new conditions of use

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Any patients with allogenic TPH
* Following in post-TPH with antigenemia or PCR-CMV
* CMV in blood test detected by antigenemia or PCR before the day 180 post-TPH
* The beginning of treatment must be Duch early as possible. Maximum in the 72 hours from the antigenemia or PCR-CMV detection
* Be the first or second time of a CMV infection
* Sign the informed consent
* Pregnancy negative test in fertile age patients

Exclusion Criteria:

* Patients received auto or syngenic TPH
* Patients <50 kg weight
* Known allergy or hypersensibility patients to valganciclovir, ganciclovir or aciclovir
* Digestive intolerant: nauseous, vomit and or diarrhea that could difficult oral administration of valganciclovir
* Patients that presents CMV infection or that is being evaluated for suspected CMV
* Patients that have presented >2 CMV infection episode, before the current one
* Severe liver disease defined by bilirubin ≥ 10mg/dL
* Treated with: foscarnet, ganciclovir, cidofovir or another antiviral drug active to CMV, in the previous 30 days at the current episode
* Neutrophils < 500 /µL at the beginning of valganciclovir treatment. Patients with >500 PMN/µL and < 1000/µL must start a G-CSF treatment to get neutrophils value > 1000/µL
* Platelets < 25/mm3 even receiving transfusion
* Clearance Creatinine < 10mL/min or dialysed patients
* Pregnancy or lactant women
* Other contraindication detailed in the "filling card"
* Previous inclusión in this study at the treated group. Is allowed that a patient participate as a control case and after that receive valganciclovir treatment in after CMV episode

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2005-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
To value valganciclovir efficacy in advance treatment of CMV in patients received allogenic transplant with a uniform treatment. | 1 year

SECONDARY OUTCOMES:
To value valganciclovir security in advance treatment of CMV in in patients received allogenic transplant with a uniform treatment. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: de la Cámara Rafael, Dr, Study Chair — Hospital Universitario La Princesa
Locations (8):
- Spain (8):
  - Hospital Clínico y Provincial de Barcelona, Barcelona, Barcelona
  - Hospital Universitario "Germans Trias i Pujol", Barcelona, Barcelona
  - Hospital Universitario de la Princesa, Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Madrid
  - Hospital Universitario Morales Meseguer, Murcia, Murcia, Murcia
  - Hospital general de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitario La Paz, Madrid
  - Hospital Clínico Universitario de Salamanca, Salamanca

REFERENCES:
- [Background] Ljungman P, Reusser P, de la Camara R, Einsele H, Engelhard D, Ribaud P, Ward K; European Group for Blood and Marrow Transplantation. Management of CMV infections: recommendations from the infectious diseases working party of the EBMT. Bone Marrow Transplant. 2004 Jun;33(11):1075-81. doi: 10.1038/sj.bmt.1704505. No abstract available. PMID 15077131
- [Background] Ljungman P, de La Camara R, Milpied N, Volin L, Russell CA, Crisp A, Webster A; Valacyclovir International Bone Marrow Transplant Study Group. Randomized study of valacyclovir as prophylaxis against cytomegalovirus reactivation in recipients of allogeneic bone marrow transplants. Blood. 2002 Apr 15;99(8):3050-6. doi: 10.1182/blood.v99.8.3050. PMID 11929799
- [Background] Reusser P, Einsele H, Lee J, Volin L, Rovira M, Engelhard D, Finke J, Cordonnier C, Link H, Ljungman P; Infectious Diseases Working Party of the European Group for Blood and Marrow Transplantation. Randomized multicenter trial of foscarnet versus ganciclovir for preemptive therapy of cytomegalovirus infection after allogeneic stem cell transplantation. Blood. 2002 Feb 15;99(4):1159-64. doi: 10.1182/blood.v99.4.1159. PMID 11830461
- [Background] Razonable RR, Paya CV. Valganciclovir for the prevention and treatment of cytomegalovirus disease in immunocompromised hosts. Expert Rev Anti Infect Ther. 2004 Feb;2(1):27-41. doi: 10.1586/14787210.2.1.27. PMID 15482169
- [Background] Cvetkovic RS, Wellington K. Valganciclovir: a review of its use in the management of CMV infection and disease in immunocompromised patients. Drugs. 2005;65(6):859-78. doi: 10.2165/00003495-200565060-00012. PMID 15819597
- [Background] Paya C, Humar A, Dominguez E, Washburn K, Blumberg E, Alexander B, Freeman R, Heaton N, Pescovitz MD; Valganciclovir Solid Organ Transplant Study Group. Efficacy and safety of valganciclovir vs. oral ganciclovir for prevention of cytomegalovirus disease in solid organ transplant recipients. Am J Transplant. 2004 Apr;4(4):611-20. doi: 10.1111/j.1600-6143.2004.00382.x. PMID 15023154
- [Background] Clark BS, Chang IF, Karpen SJ, Herrera L, Scott JD, Bristow LJ, Quiros-Tejeira RE, Goss JA. Valganciclovir for the prophylaxis of cytomegalovirus disease in pediatric liver transplant recipients. Transplantation. 2004 May 15;77(9):1480. doi: 10.1097/01.tp.0000123081.81022.33. No abstract available. PMID 15167619
- [Background] Ciancio G, Burke GW, Mattiazzi A, Leibovici Z, Dowdy L, Roth D, Kupin W, Rosen A, Jorge D, Cirocco RE, Miller J. Cytomegalovirus prophylaxis with valganciclovir in kidney, pancreas-kidney, and pancreas transplantation. Clin Transplant. 2004 Aug;18(4):402-6. doi: 10.1111/j.1399-0012.2004.00180.x. PMID 15233817
- [Background] Einsele H, Reusser P, Hertenstein B, Bornhäuser M, Kröger N, Kahls P, et al. Pharmakokinetics of Valganciclovir after AlloSCT: A Fixed Oral Dose Can Be Used for Preemptive Therapy in Patients with Normal Body Weight - Even with Intestinal GVHD. Blood 2004;104(11):abstract 2239.
- [Background] Ljungman P, Griffiths P, Paya C. Definitions of cytomegalovirus infection and disease in transplant recipients. Clin Infect Dis. 2002 Apr 15;34(8):1094-7. doi: 10.1086/339329. Epub 2002 Mar 11. PMID 11914998
- [Background] Burri M, Wiltshire H, Kahlert C, Wouters G, Rudin C. Oral valganciclovir in children: single dose pharmacokinetics in a six-year-old girl. Pediatr Infect Dis J. 2004 Mar;23(3):263-6. doi: 10.1097/01.inf.0000116760.16582.a9. PMID 15014306
- [Background] Nichols WG, Corey L, Gooley T, Drew WL, Miner R, Huang M, Davis C, Boeckh M. Rising pp65 antigenemia during preemptive anticytomegalovirus therapy after allogeneic hematopoietic stem cell transplantation: risk factors, correlation with DNA load, and outcomes. Blood. 2001 Feb 15;97(4):867-74. doi: 10.1182/blood.v97.4.867. PMID 11159510
- See also: Spanish association of Haematology — http://www.aehh.org